CLINICAL TRIAL: NCT06542978
Title: Effect of Prophylactic Application of 40Hz Transcranial Stimulation in AICU on Incidence of Postoperative Delirium in Elderly Patients Undergoing Elective Gastrointestinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Henan FYX
Record Dates: First submitted 2024-07-23; First posted 2024-08-07 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Delirium; Anesthesia; Elderly
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40Hz stimulation group (Experimental): After admission to AICU, the experimental group was stimulated at 40Hz for 6h;
  Interventions: Device: 40Hz stimulation
- Control group (No Intervention): After admission to AICU, the control group was not stimulated at 40Hz ;

INTERVENTIONS:
Device: 40Hz stimulation — Exogenous 40HZ stimulation is a physical intervention that can drive oscillations in the gamma range, and the oscillations and pulses caused at the corresponding frequency can lead to a significant reduction in β-amyloid, reverse tau hyperphosphorylation, and thereby improve the cognitive function of patients.
  Arms: 40Hz stimulation group

SUMMARY:
Postoperative delirium is an acute central nervous system dysfunction caused by surgical stress, which is manifested by postoperative acute, non-specific changes in consciousness level, attention, cognitive ability and disturbance of sleep and wake cycles. It is one of the most common surgical complications in the elderly, occurring in more than 75% of patients receiving mechanical ventilation in the intensive care unit(ICU).Exogenous 40 Hz stimulation can improve cognitive functioning.Therefore, the aim of this study was to investigate the effect of exogenous 40Hz stimulation on the incidence of postoperative delirium in elderly patients undergoing elective gastrointestinal surgery in AICU.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 65 years old,gender not limited
* 2.ASA classification Ⅱ ~ Ⅳ
* 3.Elective gastrointestinal general anesthesia surgery

Exclusion Criteria:

* 1.History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis
* 2.Pre-operative coma, severe dementia, speech impairment or severe illness incapacitated and unable to communicate
* 3.Delirium on admission or pre-operative delirium, brain injury
* 4.Severely infected person
* 5.Severe liver dysfunction (Child-Pugh C), severe renal insufficiency (preoperative dialysis)
* 6.Severe hearing or vision impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Day 1, Day 2, Day 3 ,Day 4, Day 5, Day 6,Day 7 after surgery
  Postoperative delirium was assessed using the CAM-ICU scale.The RASS score (The Richmond Agitation-Sedation Scale) was used to assess arousal. When the patient's RASS score is not -4 /-5, delirium evaluation can continue considering the patient's wakefulness status.CAM-ICU scale contains four features (Feature 1, Feature 2, Feature 3, and Feature 4). Delirium can be diagnosed when the patient is positive for features 1, 2, 3, or 4.

SECONDARY OUTCOMES:
Blood Markers | half hour, 6hours, 24hours and 48hours after transfer to aicu
  Serum Tau proteomic analysis and CRP, IL-6, and TNF-ɑ were recorded
Sleep quality | 8:00 to 10:00 every morning for the first three days after surgery
  The Chinese version of the Richards-Campbell Sleep Quality Scale Score (RCSQ) was used to evaluate sleep quality. RCSQ scoring average for five projects, including 0 ~ 25 points on behalf of the poor quality of sleep, on behalf of the sleep quality of 76 ~ 100 points; The higher the score says sleep quality, the better
The incidence of pain | 6hours, 24hours, 48hours after surgery
  Mark a 0-10cm horizontal line on the paper with a ruler, and determine the score in millimeters (mm). The score range is 0-100mm, and the higher the score, the greater the pain intensity; No pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), severe pain (75-100 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Henan People's Hospital, Zhengzhou, Henan, China